CLINICAL TRIAL: NCT01481311
Title: Detection of Patients With Abnormal Water Distribution Based on Bioelectrical Impedance Analysis (BIA)
Status: Completed | Type: Observational
Sponsor: Seca GmbH & Co. Kg. (Industry)
Responsible Party: Sponsor
Other Study IDs: BCA-05
Record Dates: First submitted 2011-11-10; First posted 2011-11-29 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Deuterium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients before dialysis treatment
  Interventions: Device: medical Body Composition Analyzer seca 514/515; Procedure: Deuterium and Sodium Bromide dilution methods
- Patients after dialysis treatment
  Interventions: Device: medical Body Composition Analyzer seca 514/515; Procedure: Deuterium and Sodium Bromide dilution methods

INTERVENTIONS:
Device: medical Body Composition Analyzer seca 514/515 — Current of 100 µA
Procedure: Deuterium and Sodium Bromide dilution methods — Orally administered to the subject in a solution with 100 ml tap water.

SUMMARY:
The aim of this clinical investigation is to prove that the seca mbca detects dialysis patients with abnormal water distribution correctly. Abnormal high water distribution is defined as more than 2 liters of Total Body Water (TBW) above a normal value range. TBW and Extra Cellular Water (ECW) are calculated with prediction equations for healthy subjects generated in BCA-01. The results are compared with TBW and ECW ascertained by dilution methods as standard reference methods. The Bioelectrical Impedance Analysis (BIA) method should be evaluated to the accuracy of the absolute measurement of the volume state of dialysis patients (euvolaemic and hypervolaemic) based on a single measurement.

ELIGIBILITY:
Inclusion Criteria:

The study will cover 50 adults. Men and women in an age range of 18 to 65 years and a Body Mass Index (BMI) range of 18.5 to 35 kg/m2 should be equally distributed. Subjects have to be patients with chronic kidney failure taking dialysis treatment. 25 patients are taken before and another 25 patients after this treatment. Patients that are taken before dialysis treatment should have been dialysed two and not three days before.

Exclusion Criteria:

* amputation of limbs
* gastrointestinal tract illnesses that influence the absorption of substances that are needed for dialysis
* bed-ridden patients patients with clinical relevant hypervolaemia or hypovolaemia
* electrical implant as cardiac pacemaker
* insulin pumps
* pregnancy or breastfeeding period
* subjects who cannot provide an Informed Consent Form (ICF) by themselves
* subjects who might be dependent from the sponsor or the investigation site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of 50 patients suffering from kidney disease are planned to be collected.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Bioelectrical impedance (Resistance and Reactance) of 5 and 50 kHz for the right body side | about 2 minutes
  The measurements are utilized as input for prediction equations to calculate TBW and ECW.

SECONDARY OUTCOMES:
Bioelectrical impedance (Resistance and Reactance) of 1, 1.5, 2, 3, 7.5, 10, 15, 20, 30, 75, 100, 150, 200, 300, 500, 750 and 1,000 kHz | about 2 minutes
  The measurement is planned to be done for all body segments: right arm, left arm, right leg, left leg, trunk, right body side and left body side. In total resistance and reactance at 19 frequencies for 7 body segments are to be measured.
TBW | within 4 hours
  A D2O dose of 400 mg per kg body weight mixed with tap water is administered orally in the morning fasting and after a 2 hour fluid abstention. The distribution of the stable isotope in the TBW is completed after 4 hours. During this period, the subject remains fasting. Two venous blood samples of 10 ml whole blood are taken immediately before and four hours after taking D2O. The plasma samples are analyzed using Isoptopic Ratio Mass Spectrometry (IRMS).
ECW | within 4 hours
  Orally administered NaBr is resorbed quickly and completely and almost exclusively distributes in the extracellular compartment. Blood samples of 10 ml are taken immediately before and 4 hours after oral application of 50 mg NaBr per kg body weight. The serum sample is analyzed by X-Ray Fluorescence Spectroscopy (XRF).

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Slowinski, Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité University Medicine Berlin, Berlin, State of Berlin, Germany